CLINICAL TRIAL: NCT07300202
Title: CLINICAL RESEARCH PROTOCOL [A Phase I, Single-arm, Open-label, Dose-escalation Clinical Study to Evaluate the Safety and Tolerability of Orialpha (BD-C) in Healthy Adult Volunteers]
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oriplantee Company Limited (Other)
Collaborators: Vietstar Biomedical Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORIPLANTEE
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Evaluate the Safety Profile and Tolerability of Orialpha in Healthy Adult Volunteers; Breast Cancer
Keywords: Orialpha; breast cancer; phase 1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, dose-escalation study using a traditional 3+3 design. Healthy adult volunteers will be enrolled sequentially into five ascending dose cohorts: 0.25×, 0.5×, 1×, 1.5×, and 2× the anticipated dose. Safety and tolerability will be assessed after each cohort prior to escalation to the next dose level. All participants will receive the investigational product, Orialpha (BD-C), and there is no comparator or placebo group
Masking Description: No blinding is performed. This is an open-label study in which participants, investigators, and study staff are aware of the investigational product being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm - Orialpha (BD-C) (Experimental): Participants in this single-arm, open-label, dose-escalation study will sequentially receive ascending doses of the investigational product Orialpha (BD-C) according to a traditional 3+3 design. The five planned dose levels are:
  0.25× anticipated dose
  0.5× anticipated dose
  1. anticipated dose
     1.5× anticipated dose
  2. anticipated dose Safety and tolerability will be assessed after each cohort before escalating to the next dose level. All participants receive the investigational product; there is no comparator or placebo group.
  Interventions: Drug: Orialpha (BD-C)

INTERVENTIONS:
Drug: Orialpha (BD-C) — Orialpha (BD-C) is a botanical investigational product derived from Uvaria grandiflora (Bù dẻ tía), with Zeylenone as its primary active compound. Participants will receive a single dose according to the assigned dose cohort. Safety, tolerability, and maximum tolerated dose (MTD) will be evaluated sequentially following the traditional 3+3 dose-escalation design.

SUMMARY:
This Phase I clinical study is designed to evaluate the safety and determine the maximum tolerated dose (MTD) of Orialpha (BD-C) in healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase I, single-arm, open-label, dose-escalation clinical study is designed to evaluate the safety and determine the maximum tolerated dose (MTD) of Orialpha (BD-C) in healthy adult volunteers. The study aims to:

* Determine the frequency and severity of treatment-related adverse events, adverse events leading to discontinuation, and serious adverse events (SAEs) within each cohort.
* Assess the effects of Orialpha on hematology and biochemistry parameters before dosing and after the final dose in each cohort.

Healthy volunteers who meet all eligibility criteria will receive the investigational product for 7 days. The first cohort will include 3 participants receiving the lowest dose (0.25 × the anticipated clinical dose). Following safety evaluation, subsequent cohorts will receive higher dose levels (0.5 ×, 1.0 ×, 1.5 ×, and 2.0 × the anticipated clinical dose) according to predefined dose-escalation rules.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, aged 18 to 60 years.
2. No clinically significant abnormalities in hematology, biochemistry, electrocardiogram (ECG), or vital signs as assessed by the investigator.
3. Willing to voluntarily participate in the study by signing the informed consent form.
4. Able to comply with study procedures and treatment as assessed by the investigator.

Exclusion Criteria:

1. History of allergy to herbal-derived drugs similar to the investigational product or any excipient.
2. Current or prior participation in another clinical trial involving an investigational product within the past 4 months.
3. Use of immunosuppressive drugs within 28 days prior to the first dose of Orialpha.
4. Active autoimmune disease or documented history of autoimmune disease within the past 2 years.
5. History of primary immunodeficiency.
6. Presence of any acute or chronic illness requiring treatment.
7. Inability to comply with study procedures or investigational product administration as assessed by the investigator.
8. Female subjects who are pregnant or breastfeeding, or male or female subjects of reproductive potential not using effective contraception.
9. Any condition which, in the opinion of the investigator, would interfere with the evaluation of the investigational treatment, patient safety, or interpretation of study results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Absolute number of subjects experiencing treatment-related adverse events in each cohort | From the first dose administration until the final study visit (up to 90 days).
  Percentage (%) is calculated as the absolute number of treatment-related adverse events divided by the total number of subjects in the SS.
Absolute number of subjects experiencing adverse events leading to study discontinuation in each cohort | From the first dose administration until the final study visit (up to 90 days)
  Percentage (%) is calculated as the absolute number of adverse events leading to discontinuation divided by the total number of subjects in the SS.
Absolute number of subjects experiencing serious adverse events (SAEs) in each cohort | From the first dose administration until the final study visit (up to 90 days).
  Percentage (%) is calculated as the absolute number of SAEs divided by the total number of subjects in the SS

SECONDARY OUTCOMES:
Biochemistry and hematology test values (quantitative variables) before and after the study | Compared between Screening Visit (V0) and End of Treatment Visit (V2), approximately 7 days apart
  The variables will be presented in a shift table with three categories: "normal," "abnormal - not clinically significant," and "abnormal - clinically significant" at both pre-study and post-study time points.
  A summary of laboratory parameters will be described in accordance with US FDA requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No